CLINICAL TRIAL: NCT00929240
Title: A Randomized Study of the Effect of Maintenance Therapy With Bevacizumab + Capecitabine Versus Bevacizumab Alone on Progression-free Survival in Patients With HER2-negative Metastatic Breast Cancer That Has Not Progressed During First-line Docetaxel Plus Bevacizumab Therapy
Brief Title: A Study of Avastin (Bevacizumab) + Xeloda (Capecitabine)as Maintenance Therapy in Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22223; 2008-006872-31
Record Dates: First submitted 2009-06-16; First posted 2009-06-26 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Capecitabine

ARMS (2):
- Avastin (bevacizumab) (Active Comparator)
  Interventions: Drug: bevacizumab [Avastin]
- Avastin (bevacizumab) + Xeloda (capecitabine) (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15 mg/kg iv on day 1 of each 3 week cycle (maintenance phase)
Drug: capecitabine [Xeloda] — 1000 mg/m2 po bid on days 1-14 of each 3 week cycle (maintenance phase)
  Arms: Avastin (bevacizumab) + Xeloda (capecitabine)

SUMMARY:
This randomized study will compare maintenance therapy with Avastin (bevacizumab) + Xeloda (capecitabine) versus Avastin alone, in patients with HER2-negative metastatic breast cancer who have not progressed during first-line therapy with docetaxel + Avastin. Eligible patients will receive up to 6 x 3 week cycles of treatment with Avastin (15 mg/mg IV on Day 1 of each cycle) + docetaxel (75-100 mg/m2 IV on Day 1 of each cycle). Those patients who do not progress will be randomized to 3 week cycles of either a) Avastin (15 mg/kg IV on Day 1 of each cycle) + Xeloda (1000 mg/m2 po bid on Days 1-14 of each cycle) or b) Avastin alone. Study treatment will continue until disease progression, unacceptable toxicity, patient request for withdrawal or end of study, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* HER2-negative metastatic breast cancer
* candidates for taxane-based chemotherapy;
* ECOG performance status of 0 or 1.

Exclusion Criteria:

* previous chemotherapy for metastatic breast cancer;
* prior adjuvant/neo-adjuvant chemotherapy within 6 months prior to study;
* prior radiotherapy for treatment of metastatic disease;
* chronic daily treatment with aspirin (325 mg/day) or clopidogrel(>75mg/day).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- Brazil (8):
  - Fortaleza, Ceará
  - Belo Horizonte, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Ijuí, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Jaú, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
- China (3):
  - Beijing
  - Hangzhou
  - Shanghai
- Egypt (2):
  - Alexandria
  - Cairo
- France (13):
  - Amiens
  - Angers
  - Besançon
  - Bobigny
  - Dijon
  - Hyères
  - Le Coudray
  - Lille
  - Paris
  - Périgueux
  - Rodez
  - Saint-Priest-en-Jarez
  - Strasbourg
- Hong Kong, Hong Kong
- India (4):
  - Bangalore
  - Hyderabad
  - Mumbai
  - New Delhi
- Italy (6):
  - Brindisi, Apulia
  - Napoli, Campania
  - Trieste, Friuli Venezia Giulia
  - Genoa, Liguria
  - Saronno, Lombardy
  - Antella (FI), Tuscany
- Poland (2):
  - Bydgoszcz
  - Wroclaw
- Saudi Arabia (2):
  - Dammam
  - Jeddah
- Spain (8):
  - Alcoy, Alicante
  - Sabadell, Barcelona, Barcelona
  - Alcazar de S. Juan, Ciudad Real
  - Jaén, Jaen
  - Málaga, Malaga
  - Toledo, Toledo
  - Valencia, Valencia
  - Barakaldo, Vizcaya
- Turkey (Türkiye) (4):
  - Ankara
  - Antalya
  - Istanbul
  - Sıhhiye, Ankara

REFERENCES:
- [Derived] Gligorov J, Doval D, Bines J, Alba E, Cortes P, Pierga JY, Gupta V, Costa R, Srock S, de Ducla S, Freudensprung U, Mustacchi G. Maintenance capecitabine and bevacizumab versus bevacizumab alone after initial first-line bevacizumab and docetaxel for patients with HER2-negative metastatic breast cancer (IMELDA): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1351-60. doi: 10.1016/S1470-2045(14)70444-9. Epub 2014 Sep 28. PMID 25273343

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Treatment Phase: Bevacizumab Plus (+) Docetaxel: During the Initial Phase all participants received bevacizumab 15 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first. Participants also received docetaxel, a recommended dose of 100 milligrams per square meter (mg/m^2) IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Treatment Phase, participants with an objective response (PR or CR) or SD following 3-6 cycles of bevacizumab + docetaxel were randomized to receive maintenance therapy with either bevacizumab alone or bevacizumab + capecitabine.
- Maintenance Phase: Bevacizumab: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first along with docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Phase, participants with an objective response (partial response [PR] or complete response [CR]) or disease stabilization (SD) received 15 mg/kg bevacizumab IV on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, participant request for withdrawal or end of study, whichever occurred first.
- Maintenance Phase: Bevacizumab + Capecitabine: During the Initial Phase participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or withdrawal, whichever occurred first, along with docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Phase, participants with an objective response were randomized to receive bevacizumab 15 mg/kg IV on Day 1 of each 3-week cycle plus capecitabine 1000 mg/m^2 twice daily on Days 1 to 14 of each 3 week cycle until disease progression, unacceptable toxicity, request for withdrawal or end of study, whichever occurred first. If one of the drugs was discontinued before disease progression, treatment was continued with the second drug until disease progression, unacceptable toxicity, withdrawal or end of study, whichever occurred first.
Period: Initial Treatment Phase
Arm/Group | Initial Treatment Phase: Bevacizumab Plus (+) Docetaxel | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Started | 284 (Includes only the participants that received Initial Phase Treatment.) | 0 (Participants were randomized to 1 of 2 treatment groups at the end of the initial treatment phase.) | 0
Completed | 185 (Participants were randomized to 1 of 2 treatment groups at the end of the initial treatment phase.) | 0 | 0
Not Completed | 99 | 0 | 0
Not completed — Adverse Event | 31 | 0 | 0
Not completed — Disease progression | 41 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Health authority/Study termination | 3 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Period: Maintenance Phase
Arm/Group | Initial Treatment Phase: Bevacizumab Plus (+) Docetaxel | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Started | 0 (Participants were randomized to 1 of 2 treatment groups at the end of the initial treatment phase.) | 94 | 91
Completed | 0 | 0 | 0
Not Completed | 0 | 94 | 91
Not completed — Disease progression | 0 | 73 | 60
Not completed — Adverse Event | 0 | 9 | 12
Not completed — Withdrawal by Subject | 0 | 2 | 6
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Health authority/Study termination | 0 | 1 | 2
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Change of treatment | 0 | 4 | 0
Not completed — Treatment ongoing at study closure | 0 | 0 | 10
Not completed — Participant not treated | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Initial Phase Intent-to-Treat (ITT) population: all participants who were enrolled.
Groups:
- Intial Treatment Phase: Bevacizumab + Docetaxel: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first. Participants also received docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Treatment Phase, participants with an objective response (PR or CR) or SD following 3-6 cycles of bevacizumab + docetaxel were randomized to receive maintenance therapy with either bevacizumab alone or bevacizumab + capecitabine.
Arm/Group | Intial Treatment Phase: Bevacizumab + Docetaxel
Number analyzed (Participants) | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death (Maintenance Phase Data Cutoff October 4, 2013)
Description: Progression Free Survival (PFS) was defined as the time from first study drug dosing (during the maintenance treatment phase) to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST). Progressive Disease (PD) was defined as a 20 percent (%) or greater increase in the sum of the Longest Diameter (LD) of the target lesions taking as reference the smallest sum LD recorded or appearance of new lesions.
Time Frame: Randomization, at the end of every third cycle (every 9 weeks) until the end of maintenance phase and every 3 months until disease progression or death until data cutoff on October 4, 2013, up to 4 years
Population: Maintenance Phase ITT population: All randomized participants
Measure: Number; unit: percentage of participants
Groups:
- Maintenance Phase: Bevacizumab: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first along with docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Phase, participants with an objective response (PR or CR) or SD received 15 mg/kg bevacizumab IV on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, participant request for withdrawal or end of study, whichever occurred first.
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants | 88.3 | 75.8

2. Primary Outcome: Progression Free Survival (Maintenance Phase Data Cutoff October 4, 2013)
Description: PFS was defined as the time from first study drug dosing to the first documented disease progression or death, whichever occurred first.Time to progression was defined as the time from randomization to the first documented disease progression defined per RECIST 1.0 criteria. Participants without an event at data cut-off or who were withdrawn from the study without documented progression were censored at the date of the last tumor assessment when the participant was known to be progression free. Participants who took other non-protocol anti-cancer drugs while being on study medication, and who were still event free were censored on the date of first dose of the anti-cancer drug. Participants without post-randomization tumor assessments but alive were censored at the time of randomization. Participants without post-randomization assessments, who died after randomization were considered to have the PFS event at date of death. Kaplan-Meier estimation was used for median time to PFS
Time Frame: as for outcome 1
Population: Maintenance Phase ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
months | 4.3 [3.9 to 6.8] | 11.9 [9.8 to 15.4]
Statistical Analysis 1: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p < 0.0001, Log Rank — Stratified by interactive voice/Web response system (IVRS), estrogen receptor (ER) status, visceral metastasis (yes/no), response to initial phase, and lactate dehydrogenase (LDH) level; Hazard Ratio (HR) = 0.383, 95% CI 2-sided [0.266 to 0.551] — Stratified by IVRS, ER status, visceral metastasis (yes/no), response to initial phase, and LDH level
Statistical Analysis 2: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p < 0.0001, Log Rank; Unstratified analysis; Hazard Ratio (HR) = 0.429, 95% CI 2-sided [0.309 to 0.597]

3. Secondary Outcome: Percentage of Participants With Best Overall Confirmed Objective Response of CR or PR Per RECIST 1.0 (Maintenance Phase Data Cutoff October 4, 2013)
Description: Objective Response was determined by the investigator using modified RECIST criteria, Version 1.0. An objective response was a complete or partial overall confirmed response as determined by investigators. CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as greater than or equal to (≥) 30 % decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. Progressive disease (PD) was defined as 20% increase in the sum of the longest diameter of target lesions and SD was defined as small changes that do not meet above criteria. Pearson-Clopper one-sample method was used for Confidence intervals (CIs).
Time Frame: as for outcome 1
Population: Maintenance Phase ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants | 76.6 [66.7 to 84.7] | 85.7 [76.8 to 92.2]
Statistical Analysis 1: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p = 0.113, Chi-squared; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [-2.1 to 20.3] — CIs with Hauck-Anderson adjustment for difference in rates of bevacizumab + capecitabine arm to bevacizumab alone arm

4. Secondary Outcome: Percentage of Participants With Clinical Benefit (CR, PR and SD) Per RECIST 1.0 (Data Cutoff October 4, 2013)
Description: CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as ≥ 30 % decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. SD was defined as small changes that do not meet above criteria.
Time Frame: as for outcome 1
Population: Maintenance Phase ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants | 97.9 [92.5 to 99.7] | 98.9 [94.0 to 100.0]
Statistical Analysis 1: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p = 0.580, Chi-squared; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.6 to 4.6] — CIs with Hauck-Anderson adjustment for difference in rates of Bevacizumab+Capecitabine group to Bevacizumab only group

5. Secondary Outcome: Percentage of Participants Who Died (Maintenance Phase Data Cutoff October 4, 2013)
Time Frame: as for outcome 1
Population: Maintenance Phase ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants | 56.4 | 36.3

6. Secondary Outcome: Overall Survival (Maintenance Phase Data Cutoff October 4, 2013)
Description: Duration of Overall Survival (OS) was defined as the time from randomization to death of any cause. The OS data for participants for whom no death was captured in the clinical database were censored at the last time they were known to be alive. Kaplan Meier estimation was used to determine OS.
Time Frame: as for outcome 1
Population: Maintenance Phase ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
months | 23.7 [18.5 to 31.7] | 39.0 [32.3 to NA] — Upper Confidence limit was not estimated because of the large number of censored events.
Statistical Analysis 1: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p < 0.0003, Log Rank — Stratified by IVRS, ER status, visceral metastasis (yes/no), response to initial phase, and LDH level; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.263 to 0.685]
Statistical Analysis 2: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p = 0.002, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 0.516, 95% CI 2-sided [0.334 to 0.798]

7. Secondary Outcome: Percentage of Participants Expected to Be Alive After 1 and 2 Years on Treatment (Maintenance Phase Data Cutoff October 4, 2013)
Description: Probability of being alive after 1 and 2 years on treatment with 95% CIs was calculated using Kaplan Meier approach with LOGLOG transformation.
Time Frame: Years 1 and 2
Population: Maintenance Phase ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants
  1 Year | 71.6 [61.1 to 79.7] | 90.4 [81.8 to 95.1]
  2 Years | 49.4 [38.5 to 59.3] | 69.0 [57.6 to 77.9]

8. Secondary Outcome: Percentage Of Participants With PD or Death Due to PD (Maintenance Phase Data Cutoff October 4, 2013)
Description: PD was defined per RECIST 1.0 as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Randomization, at the end of every third cycle (every 9 weeks) until the end of maintenance phase and every 3 months until disease progression or death until data cutoff on October 4, 2013
Population: Maintenance Phase ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
percentage of participants | 88.3 | 74.7

9. Secondary Outcome: Time To Progression (Maintenance Phase Data Cutoff October 4, 2013)
Description: Time to Progression was defined as the time from randomization to the first documented disease progression (using investigator assessments of disease progression by RECIST 1.0). PD was defined as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: as for outcome 8
Population: Maintenance Phase ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 94 | 91
months | 4.3 [3.9 to 6.8] | 11.9 [9.8 to 15.4]
Statistical Analysis 1: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p < 0.0001, Log Rank — Stratified by IVRS, ER status, visceral metastasis (yes/no), response to initial phase, and LDH level; Hazard Ratio (HR) = 0.383, 95% CI 2-sided [0.266 to 0.551] — Stratification variables are randomisation stratification parameters as of IVRS: ER status, Visceral metastasis (yes/no), Response to initial phase, LDH concentration level
Statistical Analysis 2: Comparison: Maintenance Phase: Bevacizumab vs Maintenance Phase: Bevacizumab + Capecitabine; Test type: Superiority or Other; p < 0.0001, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.305 to 0.591] — Hazard ratio was determined using the cox regression model

10. Secondary Outcome: Quality of Life Assessed As Change From Baseline in Global Health Status Using The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - 30 (EORTC QLQ - C30) (Maintenance Phase Data Cutoff October 4, 2013)
Description: The EORTC QLQ-C30 incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnoea, insomnia, appetite loss, constipation, diarrhea and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores were averaged and transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms. The change in global health status was determined to be the difference in values at baseline and each specific visit. The term ''baseline'' refers to the time of randomization to the maintenance phase.
Time Frame: Baseline, Randomization and Cycles 3, 6, 9 and 12
Population: Maintenance Phase ITT population; n (number) = number of participants analyzed at the specific visit. Only timepoints with more than 10 participants in each treatment arm are presented.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Maintenance Phase: Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Number analyzed (Participants) | 83 | 86
units on a scale
  Randomization (n= 83, 86) | -3.51 [-9.63 to 2.60] | -4.46 [-9.40 to 0.48]
  Cycle 3 (n= 44, 52) | 0.76 [-6.65 to 8.17] | -3.21 [-9.99 to 3.58]
  Cycle 6 (n= 26, 54) | 4.17 [-6.49 to 14.82] | -5.40 [-11.67 to 0.87]
  Cycle 9 (n= 18, 37) | 8.80 [-4.57 to 22.17] | -1.80 [-8.92 to 5.32]
  Cycle 12 (n= 12, 31) | 0.69 [-17.99 to 19.37] | 0.00 [-8.24 to 8.24]

11. Secondary Outcome: Percentage of Participants With Best Overall Confirmed Objective Response of CR or PR Per RECIST 1.0 (Initial Treatment Phase)
Description: Objective Response was determined by the investigator using RECIST criteria, Version 1.0. An objective response was a complete or partial overall confirmed response as determined by investigators. CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as ≥ 30% decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. Pearson-Clopper one-sample method was used for CI.
Time Frame: Screening and at the end of every third cycle until randomization for an average of 18 weeks
Population: Initial Phase ITT population; only participants who were not randomized at the end of the initial treatment phase were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Initial Treatment Phase: Bevacizumab + Docetaxel: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first, along with docetaxel a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion.At the end of the Initial Treatment Phase, participants with an objective response (PR or CR) or SD following 3-6 cycles of bevacizumab + docetaxel were randomized to receive maintenance therapy with either bevacizumab alone or bevacizumab + capecitabine.
Arm/Group | Initial Treatment Phase: Bevacizumab + Docetaxel
Number analyzed (Participants) | 102
percentage of participants | 8.8 [4.1 to 16.1]

12. Secondary Outcome: Percentage of Participants With Clinical Benefit (CR, PR and SD) Per RECIST 1.0 (Initial Treatment Phase)
Description: CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as ≥30% decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. SD was defined as small changes that do not meet above criteria.
Time Frame: Screening and at the end of every third cycle until randomization for an average of 18 weeks
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Initial Treatment Phase: Bevacizumab + Docetaxel: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first, along with docetaxel a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Treatment Phase, participants with an objective response (PR or CR) or SD following 3-6 cycles of bevacizumab + docetaxel were randomized to receive maintenance therapy with either bevacizumab alone or bevacizumab + capecitabine.
Arm/Group | Initial Treatment Phase: Bevacizumab + Docetaxel
Number analyzed (Participants) | 102
percentage of participants | 56.9 [46.7 to 66.6]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded from the date of randomization until the end of study at the cutoff date of October 4, 2013.
Description: AEs were recorded for the Safety population (all participants who received at least one dose of study drug during the maintenance phase). Only Grade 3 and above AEs have been captured per protocol.
Groups:
- Initial Treatment Phase:Bevacizumab + Docetaxel: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first. Participants also received docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Treatment Phase, participants with an objective response (PR or CR) or SD following 3-6 cycles of bevacizumab + docetaxel were randomized to receive maintenance therapy with either bevacizumab alone or bevacizumab + capecitabine.
- Maintenance Phase:Bevacizumab: During the Initial Phase all participants received bevacizumab 15 mg/kg IV on Day 1 of each 3 week cycle for a minimum of 3 cycles and a maximum of 6 cycles or until disease progression, unacceptable toxicity or participant request for withdrawal, whichever occurred first along with docetaxel, a recommended dose of 100 mg/m^2 IV administered on Day 1 of each cycle. Doses of 75 to 100 mg/m^2 of docetaxel could be administered at investigator's discretion. At the end of the Initial Phase, participants with an objective response (PR or CR) or SD received 15 mg/kg bevacizumab IV on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, participant request for withdrawal or end of study, whichever occurred first.
Arm/Group | Initial Treatment Phase:Bevacizumab + Docetaxel | Maintenance Phase:Bevacizumab | Maintenance Phase: Bevacizumab + Capecitabine
Serious Adverse Events (participants affected / at risk) | 78/284 | 7/92 | 10/91
Other Adverse Events (participants affected / at risk) | 40/284 | 4/92 | 32/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Phase:Bevacizumab + Docetaxel (N=284) | Maintenance Phase:Bevacizumab (N=92) | Maintenance Phase: Bevacizumab + Capecitabine (N=91)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 17 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 1 | 0
Embolism arterial (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Phase:Bevacizumab + Docetaxel (N=284) | Maintenance Phase:Bevacizumab (N=92) | Maintenance Phase: Bevacizumab + Capecitabine (N=91)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 0 | 29
Neutropenia (Blood and lymphatic system disorders) | 29 | 1 | 2
Hypertension (Vascular disorders) | 5 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.